CLINICAL TRIAL: NCT05912491
Title: Static and Functional Transperineal Ultrasonography for Identification of Stress Urinary Incontinence
Brief Title: Transperineal Ultrasonography in Stress Urinary Incontinence
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Iwona Magdalena Gawron, M.D., PhD., Principal Investigator, Jagiellonian University
Other Study IDs: KBET/228/B/2010
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Stress Urinary Incontinence
Keywords: stress urinary incontinence, transperineal ultrasound
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Urinary stress incontinence (UI): Women with clinical symptoms of stress urinary incontinence
  Interventions: Diagnostic Test: Transperineal ultrasonography
- No Urinary stress incontinence (no-UI): Women without clinical symptoms of stress urinary incontinence
  Interventions: Diagnostic Test: Transperineal ultrasonography

INTERVENTIONS:
Diagnostic Test: Transperineal ultrasonography — Transperineal ultrasound (TPU) with a Voluson E6 (GE Medical systems, Milwaukee, WI, USA). The probe was oriented to coaxially visualise the pubic symphysis on one side and the anus and rectum on the other side of the 2D image. Next, 3D/4D ultrasound was performed to obtain an image in the coronal plane at the level of the arms of the levator ani muscle, showing the pubic symphysis and the anus. All measurements were performed in three states: during pelvic muscle relaxation, during Valsalva manoeuvre, and during perineal squeezing.

SUMMARY:
Pelvic organ prolapse (POP) and urinary incontinence (UI) are common female disorders. Accurate diagnosis of the aetiology of pelvic organ descent and prolapse with or without accompanying urination disorders is essential for appropriate therapeutic management. Imaging and functional urodynamic testing are being increasingly used in the diagnosis of this pathology, because precise assessment of the damage to the supporting and ligament apparatus is essential for therapeutic success. Pelvic floor ultrasound can facilitate dynamic assessment of static changes that occur during functional tests. Such assessments can provide additional insights into existing defects, which have explorative value and allow for targeted correction of damage, and may thus indirectly contribute to reduced rates of revision surgeries.

DETAILED DESCRIPTION:
Application of the ultrasound transducer to the patient's perineum can visualise three female pelvic compartments, and the images can be frozen to assess the positions of anatomical structures in relation to the pelvic bones and the pre-set planes as well as measure their mutual distances and predefined angles.

The aim of the study was to assess the utility of ultrasound in the detection of UI, particularly for establishing the most useful anatomical and functional parameters and to propose cut-off points for ultrasonographic parameters. The presence of stress urinary incontinence (SUI) requiring surgical management was the inclusion criterion. All patients underwent transperineal ultrasound (TPU) with a Voluson E6 (GE Medical systems, Milwaukee, WI, USA). The probe was oriented to coaxially visualise the pubic symphysis on one side and the anus and rectum on the other side of the 2D image. When all three compartments could not be visualised in one image, one image showing the anterior and medial compartments and another image showing the medial and posterior compartments were obtained instead. Next, 3D/4D ultrasound was performed to obtain an image in the coronal plane at the level of the arms of the levator ani muscle, showing the pubic symphysis and the anus. All measurements were performed in three states: during pelvic muscle relaxation, during Valsalva manoeuvre, and during perineal squeezing. The following quantitative parameters were assessed and compared across two arms of the study (with and without SUI):

* Bladder-symphysis distance (BSD) - measured as the distance between the urine bladder neck and the symphysis,
* Alpha angle - the angle between the axis of the proximal urethra and the x-axis of the symphysis pubis (central line),
* Beta angle - the angle between the line parallel to the proximal urethra and the line parallel to the distal axis of urethra,
* Gamma angle - the angle between the lower margin of the symphysis pubis and the urinary bladder neck),
* Retrovesical angle (RVA) - the angle between the axis of the proximal urethra and the tangent line to the lowest part of the posterior wall of the urinary bladder,
* Mean urethral diameter - the sum of the urethral diameters at three points (proximal, central, and distal parts) divided by 3.

ELIGIBILITY:
Inclusion Criteria:

* Stress Urinary Incontinence

Exclusion Criteria:

* Failure to obtain endpoint measurements due to lack of cooperation during the ultrasound examination
* Prior surgery for either UI or POP
* Pelvic tumours
* Lack of consent to participate in the study

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women hospitalised at the Clinical Department of Gynecological Oncology and Gynecology, University Hospital in Krakow, between July 2012 and July 2015, aged over 18 years. The presence of stress urinary incontinence (SUI) requiring surgical management was the inclusion criterion. The control group included patients without UI referred for surgery due to mild gynaecological disorders. Exclusion criteria included prior surgery for either UI or POP, pelvic tumours that could affect pelvic organ statics, and lack of informed consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2012-07-01 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Bladder-symphysis distance (BSD) | 36 months
  Distance in mm between the urine bladder neck and the symphysis
Alpha angle | 36 months
  Measurement of the angle in degrees between the axis of the proximal urethra and the x-axis of the symphysis pubis (central line)
Beta angle | 36 months
  Measurement of the angle in degrees between the line parallel to the proximal urethra and the line parallel to the distal axis of urethra
Gamma angle | 36 months
  Measurement of the angle in degrees between the lower margin of the symphysis pubis and the urinary bladder neck
Retrovesical angle (RVA) | 36 months
  Measurement of the angle in degrees between the axis of the proximal urethra and the tangent line to the lowest part of the posterior wall of the urinary bladder
Mean urethral diameter | 36 months
  Mean urethral diameter in mm obtained by summing the urethral diameters at three points (proximal, mid, and distal) and dividing the sum obtained by 3

CONTACTS AND LOCATIONS:
Overall Officials: Kazimierz Pitynski, Ph.D., Prof., Study Chair — Jagiellonian University

IPD SHARING:
Plan to Share IPD: No